CLINICAL TRIAL: NCT04178369
Title: The Effects of Proximal And Distal Tibiofibular Joint Manipulations on Foot Posture, Ankle Range of Motion, and Balance in Chronic Hemiplegic Individuals
Brief Title: The Effects of Proximal And Distal Tibiofibular Joint Manipulations on Foot Posture, Ankle Range of Motion, and Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, Caner Karartı, Hacettepe University, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019600
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Hemiplegia; Gait, Hemiplegic; Mobility Limitation
MeSH Terms: conditions — Hemiplegia; Gait Disorders, Neurologic; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Care Provider
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental-Study Group (Experimental): In addition to the conservative treatment of the control group, proximal and distal tibiofibular joint manipulations will be applied for 6 weeks.
  Interventions: Other: Proximal And Distal Tibiofibular Joint Manipulations
- Control Group (Active Comparator): All participants were given a 6-week-long physiotherapy and rehabilitation program based on the Bobath concept (conservative treatment) for 5 days a week, 45 minutes each.
  Interventions: Other: Bobath Treatment

INTERVENTIONS:
Other: Proximal And Distal Tibiofibular Joint Manipulations — For PTFJ, the experimental intervention will be based on previously published methods. Physiotherapist will make contact with the fibular head, extending to the popliteal fossa. The associated soft tissue will be pulled in a lateral direction until the metacarpophalangeal joint will be firmly stabilized behind the fibular head.
  For DTFJ, the experimental intervention will be conducted according to previously published methods. Physiotherapist will grasp and stabilize the distal tibia with one hand and grasp the distal fibula between the finger and thenar eminence of the other hand. The fibula will be translated posteriorly until the restrictive barrier (end range) will be engaged. Then a high-velocity, low-amplitude thrust will be applied through the fibula in a posterior-superior direction.
  Arms: Experimental-Study Group
Other: Bobath Treatment — All participants will be given a 6-week-long physiotherapy and rehabilitation program based on the Bobath concept for 5 days a week, 45 minutes each. The techniques will be applied by a physiotherapist who is specialized in Bobath concept. 35 different techniques will be used to improve the selective control and weight transfer of the pelvis in sitting, standing and supine/side lying positions. Moreover, soft tissue mobilization will be also used to relieve tension and loosen stiff tissues to provide biomechanical alignment and reduce pain.
  Arms: Control Group

SUMMARY:
Limited ankle dorsiflexion adversely affects the weight bearing capacity, increases the knee extensor moment and causes insufficient maneuvers to change the center of gravity of the body in patients with hemiplegia. While biomechanical studies emphasized the importance of proximal tibiofibular joint and distal tibiofibular joint manipulations for ankle dorsiflexion, no studies examining the effect of corrective manipulation techniques applied to these two joints on foot posture, range of motion and balance were observed.

DETAILED DESCRIPTION:
In chronic hemiplegic individuals, gait loss due to biomechanical disorders of the talocrural joint (TCJ) and subtalar joint (STJ) affects 50% of the population. Although foot posture is seen at the same rate in pronation and supination, approximately 30% of individuals have abnormal and asymmetric foot posture. In particular, foot posture in the direction of plantar flexion and inversion leads to limited ankle mobility. Loss of mobility can be caused by non-neural factors as well as neural factors such as spasticity and increased myostatic reflex. Due to long-term immobilization, negative changes are seen in the tissues such as bone, muscle, tendon and ligament and especially ankle dorsiflexion is limited. Limited ankle dorsiflexion adversely affects the weight bearing capacity, increases the knee extensor moment and causes insufficient maneuvers to change the center of gravity of the body in patients with hemiplegia. The main problem is the timing of the posterior foot plantar flexion after the first contact at the beginning of the posture phase; in the late phase, defective heel and forefoot rocker roll mechanism due to the failure of forward weight transfer. For these reasons, foot posture, ankle joint range of motion and balance are adversely affected in hemiplegic individuals. Biomechanical problems related to foot deformities in chronic hemiplegic individuals have been frequently associated with TCJ and STJ anomalies. However, in biomechanical studies, it is emphasized that proximal tibiofibular joint (PTFJ) and distal tibiofibular joint (DTFJ) have important roles in optimal ankle dorsiflexion. Although PTFJ is anatomically belonging to the knee, it is evaluated within the foot-ankle complex as a function. PTFJ makes slip movements during movement in TCJ. Limitations in PTFJ movement result in limitation of the endpoints of normal ankle joint movement and anterior pain in the ankle during weight bearing. Increased tension in the lateral ligaments due to plantar flexion and inversion anomalies and traumas of the ankle applies inferior directional traction force to the distal fibula.This leads to fibular rotation in the parasagittal plane. Anterior and inferior movement of the distal fibula causes inferior and posterior shifting of the PTFJ and the PTFJ locks. This locking restricts the movement of the entire fibula during ankle movements and leads to a limitation of dorsiflexion of TCJ. It is emphasized that ankle posture significantly affects DTFJ in addition to PTFJ. The anterior ligament of DTFJ is closely related to the anterior talofibular ligament (ATFL). Plantar flexion and inversion of the trauma or supination of the foot posture, etc. conditions increase the tension in the lateral ligaments and cause pathologies in ATFL. This situation adversely affects the anterior ligament of DTFJ, leading to instability risk in this joint and loss of dorsiflexion in TCJ. While biomechanical studies emphasized the importance of proximal tibiofibular joint and distal tibiofibular joint manipulations for ankle dorsiflexion, no studies examining the effect of corrective manipulation techniques applied to these two joints on foot posture, range of motion and balance were observed. It is thought that PTFJ and DTFJ also have an effect on the above mentioned biomechanical chain in functional deficiencies caused by foot posture in the direction of plantar flexion and inversion. Therefore, we aimed to investigate the effects of PTFJ and DTFJ manipulation techniques on foot posture, range of motion and balance parameters in chronic hemiplegic subjects.

ELIGIBILITY:
Inclusion Criteria:

* presence of chronic hemiplegia (˃6 months),
* the ability to stand on the hemiplegic leg on a 30-cm-high step-board,
* the ability to walk at least 10 m without any assistive device,
* presence of limitation in ankle passive dorsiflexion (contracture),
* the ability to understand and follow verbal commands,
* to be volunteer to participate in the study.

Exclusion Criteria:

* presence of any condition that is considered as a contraindication for mobilization (such as hypermobility, trauma, inflammation, etc.),
* presence of any visual, verbal, or cognitive defects (such as aphasia, unilateral neglect, etc.),
* having ankle sprain during the past 6 weeks,
* patients who had undergone foot-ankle surgeries,
* to receive any additional treatment within the time period of our study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-12-20 (Estimated); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
Foot Posture Index | 6 weeks
  This index will be used to evaluate foot posture. During the assessment, all individuals will be asked to stand in the position where they fell the most comfortable. Six different parameters of the foot posture will be evaluated and scored between (-2) and (+2). These six parameters will be as follows: the palpation of talus head in hindfoot with the thumb and forefinger, the slope above and beneath the lateral malleolus, calcaneal supination and pronation, domination at the talonavicular joint area in the forefoot, the structure of medial longitudinal arc, and adduction and abduction of the forefoot compared to the hindfoot. The parameters scored as 0 will be considered as neutral position, while positive values represent pronation, and negative values express supination.

SECONDARY OUTCOMES:
Range of Motion | 6 weeks
  Ankle ROM will be measured in the prone position and asked to flex the knee to 90°. The central axis of a 14 in. plastic goniometer will be placed on the lateral malleolus. The stationary arm of the goniometer will be placed parallel to the lateral side of the fifth metatarsal bone. The moving arm of the goniometer will be placed parallel to the center of the fibular head, and the 3 axes will be marked with a dot. The 3 marked dots will be maintained in the same position throughout the duration of the test. One physical therapist will maintain a neutral subtalar joint position while applying force to the plantar surface of the forefoot and midfoot until further movement will be firmly restricted. The second physical therapist will confirm the neutral subtalar joint position and independently measure the ankle passive and active ROM. Measurements of ankle ROM will be repeated 3 times, with results averaged for ankle ROM data analysis.
Berg Balance Scale | 6 weeks
  Berg Balance Scale will be used to evaluate balance. Each of the 14 items of this scale will be scored between 0 to 4, where 0 indicated that the movement cannot be performed and 4 indicated that the movement is performed in the best possible way. The highest possible score on this scale is 56. High scores indicate increased postural control.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] An CM, Won JI. Effects of ankle joint mobilization with movement and weight-bearing exercise on knee strength, ankle range of motion, and gait velocity in patients with stroke: a pilot study. J Phys Ther Sci. 2016 Jan;28(2):689-94. doi: 10.1589/jpts.28.689. Epub 2016 Feb 29. PMID 27065565
- [Result] An CM, Jo SO. Effects of Talocrural Mobilization with Movement on Ankle Strength, Mobility, and Weight-Bearing Ability in Hemiplegic Patients with Chronic Stroke: A Randomized Controlled Trial. J Stroke Cerebrovasc Dis. 2017 Jan;26(1):169-176. doi: 10.1016/j.jstrokecerebrovasdis.2016.09.005. Epub 2016 Oct 17. PMID 27765557
- [Result] Kluding PM, Santos M. Effects of ankle joint mobilizations in adults poststroke: a pilot study. Arch Phys Med Rehabil. 2008 Mar;89(3):449-56. doi: 10.1016/j.apmr.2007.12.005. PMID 18295622